CLINICAL TRIAL: NCT04082663
Title: Evaluating the Effects of a Removable Dental Mouthpiece on Symptoms Associated With Parkinson's
Brief Title: Dental Appliance for Parkinson's Disease
Acronym: DAPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Gammon M Earhart, Director, Program in Physical Therapy, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201904098
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Results first posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: All participants will receive a custom-fitted dental mouthpiece and asked to wear the mouthpiece for one month.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Dental Mouthpiece (Experimental): Each participant will be fitted with a maxillary orthotic (mouthpiece). The mouthpiece is fabricated with polyvinyl ethylene acetate which is non-toxic to humans.
  Interventions: Device: Dental Mouthpiece

INTERVENTIONS:
Device: Dental Mouthpiece — Participants will complete motor tasks with and without the dental mouthpiece during the in-person baseline visit. They will also be asked to wear the mouthpiece for one month, and complete sleep and quality of life questionnaires before and after wearing the mouthpiece.

SUMMARY:
The investigators are evaluating the immediate effect of a dental mouthpiece on gait and balance among people with Parkinson disease as well as longer-term feasibility use and the effect of the mouthpiece on sleep and quality of life.

DETAILED DESCRIPTION:
The investigators are conducting a pilot study with participants who have been diagnosed with Parkinson disease recruited from the community. Participants will attend one in-person visit and be custom fitted with a dental mouthpiece. Participants will be asked to wear the mouthpiece as much as possible for one month including while sleeping and during the day, except while eating.

Participants will be asked to return for a second in-person visit to repeat gait and balance (motor) measures.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of idiopathic, typical Parkinson Disease according to the United Kingdom Brain Bank Criteria, Hoehn & Yahr stages 1-3;
* stable Parkinson disease medications for the two weeks prior to baseline visit;
* be able to walk at least 10 meters at baseline with or without an assistive device;
* have their own teeth and/or dentures;
* be willing to try to wear a mouthpiece for one month;
* are over the age of 30; and
* provide written or verbal informed consent.

Exclusion Criteria:

* pre-existing medical conditions that would inhibit full participation in the study's tasks;
* absence of any dentition;
* cognitive impairments indicated by Mini Mental Status Exam (MMSE) score of <24;
* freezing of gait which moderately or severely impacts walking; or
* current use of an oral appliance (e.g., a dental mouthpiece, retainer, or braces).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gammon M Earhart, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine Program in Physical Therapy, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lane H, Rose LE, Woodbrey M, Arghavani D, Lawrence M, Cavanaugh JT. Exploring the Effects of Using an Oral Appliance to Reduce Movement Dysfunction in an Individual With Parkinson Disease: A Single-Subject Design Study. J Neurol Phys Ther. 2017 Jan;41(1):52-58. doi: 10.1097/NPT.0000000000000160. PMID 27977521
- [Background] Potter K, Brandfass K. The Mini-Balance Evaluation Systems Test (Mini-BESTest). J Physiother. 2015 Oct;61(4):225. doi: 10.1016/j.jphys.2015.04.002. Epub 2015 Jun 1. No abstract available. PMID 26044345
- [Background] Jenkinson C, Fitzpatrick R, Peto V, Greenhall R, Hyman N. The Parkinson's Disease Questionnaire (PDQ-39): development and validation of a Parkinson's disease summary index score. Age Ageing. 1997 Sep;26(5):353-7. doi: 10.1093/ageing/26.5.353. PMID 9351479
- [Background] Trenkwalder C, Kohnen R, Hogl B, Metta V, Sixel-Doring F, Frauscher B, Hulsmann J, Martinez-Martin P, Chaudhuri KR. Parkinson's disease sleep scale--validation of the revised version PDSS-2. Mov Disord. 2011 Mar;26(4):644-52. doi: 10.1002/mds.23476. Epub 2011 Feb 10. PMID 21312275
- [Background] Moeller DR. Evaluation of a Removable Intraoral Soft Stabilization Splint for the Reduction of Headaches and Nightmares in Military PTSD Patients: A Large Case Series. J Spec Oper Med. 2013 Spring;13(1):49-54. PMID 23526322

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dental Mouthpiece
Started | 20
Completed | 13
Not Completed | 7
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dental Mouthpiece
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Movement Disorders Society - United Parkinson Disease Rating Scale III [Mean (Standard Deviation); unit: scores on a scale] — Thirty-three items on the Movement Disorders Society - United Parkinson Disease Rating Scale Part III Motor Examination are rated using five response options of 0: Normal, 1: Slight, 2: Mild, 3: Moderate, 4: Severe. The items are summed for a total score indicating overall severity of motor signs and symptoms of Parkinson's disease. The minimum score is 0 reflecting normal motor functioning and the maximum score of 132 reflecting severe motor impairment. In other words, higher scores represent worse outcomes.
  scores on a scale | 37.25 (8.67)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Gait Velocity
Description: Gait velocity will be measured while walking forwards with and without the mouthpiece
Time Frame: Baseline in-person visit
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Dental Mouthpiece
Number analyzed (Participants) | 20
m/s
  WITHOUT-Mouthpiece | 1.10 (0.24)
  WITH-Mouthpiece | 1.15 (0.22)

2. Primary Outcome: Changes in Mini-Balance Evaluation Systems Test (Mini-BESTest)
Description: Balance will be measured with the Mini-Balance Evaluation Systems Test (Mini-BESTest) with and without the mouthpiece. The assessment includes 14 items each of which is rated on a three-point scale (2: Normal, 1: Moderate, 0: Severe). The 14 item scores are summed for a total score. The range of scores is 0 to 28, and higher scores indicate better balance function.
Time Frame: Baseline in-person visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dental Mouthpiece
Number analyzed (Participants) | 20
score on a scale
  WITHOUT-Mouthpiece | 19.44 (3.58)
  WITH-Mouthpiece | 19.28 (4.06)

3. Secondary Outcome: Changes in Parkinson Disease Sleep Scale
Description: Indicators of sleep quality will be measured before and after wearing mouthpiece for one-month. The visual analog scale has 15 commonly reported symptoms associated with sleep disturbance (e.g., overall quality of nights sleep, restlessness, daytime dozing). Participants mark a cross along a 10 cm line labelled worst to best state. Items are scored by measuring the distance along each line to the intersection with the cross in centimeters. Each item score can range from 0 - symptom severe and always experienced to 10 - symptom-free. The items are summed and the maximum cumulative score is 150 (free of all symptoms).
Time Frame: Baseline and One month
Population: 2 participants missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dental Mouthpiece
Number analyzed (Participants) | 11
score on a scale
  WITHOUT-Mouthpiece at Baseline | 89.32 (29.45)
  One-Month Follow-Up | 91.68 (29.94)

4. Secondary Outcome: Changes in Parkinson Disease Questionnaire-39
Description: Quality of life will be measured before and after wearing mouthpiece for one-month. This scale has 39 questions with 5 possible answers (0 = never, 1 = Occasionally, 2 = Sometimes, 3 = Often, 4 = Always). There are eight dimensions: Mobility questions (q)1-10; Activities of Daily Living q11-16; Emotional well-being q17-22; Stigma q23-26; Social Support q27-29; Cognitive impairment q30-33; Communication q34-36; and Bodily Discomfort q37-39. Dimensions are calculated on a scale of 0 to 100, 0 is no problem at all and 100 is maximum level of a problem. The formula for scoring each dimension: (sum of scores of each question in dimension/4 (max.score per question) x nos. questions in dimension)x100. The formula for a total score (called single index) is sum of dimension scores/8.
Time Frame: Baseline and One month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dental Mouthpiece
Number analyzed (Participants) | 13
score on a scale
  WITHOUT-Mouthpiece at Baseline | 18.17 (9.22)
  One-Month Follow-Up | 17.34 (11.09)

ADVERSE EVENTS:
Time Frame: One month
Arm/Group | Dental Mouthpiece
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 8/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dental Mouthpiece (N=20)
Irritation/Discomfort from mouthpiece (Product Issues) | 7 (9) — Participants noted that the mouthpiece caused mouth irritation/discomfort.
Loose filling replaced (Surgical and medical procedures) | 1 (1) — Loose filling replaced by participant's dentist; unrelated to mouthpiece

LIMITATIONS AND CAVEATS:
High number of withdrawals leading to smaller than expected number of participants to analyze outcomes over the one month period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT04082663/Prot_SAP_000.pdf